CLINICAL TRIAL: NCT00845910
Title: A Phase II Trial of Evaluating Circulating Endothelial Cell as A Surrogate Marker for Monitoring Treatment Efficacy of Docetaxel Plus Capecitabine With Bevacizumab as First Line Treatment for Patients With Locally Recurrent and Metastatic Breast Cancer
Brief Title: A Study of Circulating Endothelial Cell as Marker for Avastin (Bevacizumab) in Combination With Docetaxel Plus Xeloda (Capecitabine) as First Line Treatment for Patients With Locally Recurrent and Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: To be confirmed
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21870
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Capecitabine; Docetaxel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: docetaxel

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 of every 3 week cycle
Drug: capecitabine [Xeloda] — 900mg/m2 po on days 1-14 of every 3 week cycle
Drug: docetaxel — 60mg/m2 iv on day 1 of every 3 week cycle

SUMMARY:
This single arm study will evaluate the correlation between circulating endothelial cell levels and treatment efficacy in patients with locally recurrent and metastatic breast cancer given first line treatment with Avastin in combination with docetaxel + Xeloda.Patients will be treated with docetaxel 60mg/m2 iv on day 1, and Xeloda 900mg/m2 po on days 1-14, of each 3 week cycle, plus Avastin 7.5 mg/kg iv on day 1 of each 3 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, 18-65 years of age;
* locally recurrent and metastatic breast cancer;
* measurable or evaluable disease;
* ECOG performance status of 0-2;
* LVEF >=50% without clinical symptoms or signs of heart failure.

Exclusion Criteria:

* unknown HER2 status, or known HER2-positive status;
* prior chemotherapy for locally recurrent or metastatic disease;
* prior adjuvant or neoadjuvant taxane therapy within 12 months prior to start of treatment;
* clinical or radiological evidence of CNS metastases;
* clinically significant cardiovascular disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Every 12 weeks

SECONDARY OUTCOMES:
Time to disease progression | Event driven
Serious adverse events | At planned visits, till disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taoyuan District